CLINICAL TRIAL: NCT07282522
Title: Investigation of Somatosensory Perception, Pain, Kinesiophobia, and Upper Extremity Functional Skills in Cervical Disc Herniation: A Case-Control Study
Brief Title: Sensory and Functional Impairments in Cervical Disc Herniation
Status: Recruiting | Type: Observational
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Dilan Demirtaş Karaoba, assistant professor, Inonu University
Other Study IDs: 2025/8426
Record Dates: First submitted 2025-12-02; First posted 2025-12-15 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Cervical Disc Herniation
MeSH Terms: interventions — Pain Threshold

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Individuals with SDH: Individuals with SDH are patients diagnosed with cervical disc herniation by a physical therapist.
  Interventions: Other: Somatosensory Perception Tests; Other: The Visual Analog Scale; Other: Pain Threshold and Tolerance Assessment; Other: Upper extremity functionality
- healthy participants.: Individuals with similar demographic characteristics who did not have any neck pain during the initial interview were considered healthy participants.
  Interventions: Other: Somatosensory Perception Tests; Other: The Visual Analog Scale; Other: Pain Threshold and Tolerance Assessment; Other: Upper extremity functionality

INTERVENTIONS:
Other: Somatosensory Perception Tests — Tactile Localization Test The tactile localization test assesses touch perception. Finger Recognition Test The participant is asked to point to their finger, which has been touched with a pen, while their eyes are closed.
  Double-Touch Stimulus Perception Test This test is based on the identification of two separate stimuli presented simultaneously.
Other: The Visual Analog Scale — The Visual Analog Scale evaluates the intensity of pain felt by patients in different activities and time periods (rest, activity and night) in centimeters (cm).
Other: Pain Threshold and Tolerance Assessment — Participants' pain threshold and tolerance to pressure are assessed using a digital algometer (JTech Medical Industries, ZEVEX Company).
Other: Upper extremity functionality — Upper extremity functionality will be assessed using the DASH and Purdue Pegboard Manual Dexterity Test.

SUMMARY:
The aim of the study was to evaluate the levels of somatosensory perception, pain threshold and kinesiophobia in individuals with SDH, to examine their relationship with upper extremity functional skills and to compare them with healthy individuals.

DETAILED DESCRIPTION:
Cervical disc herniation (SDH) occurs when nerve roots and/or spinal cord are compressed due to degeneration or displacement of the cervical intervertebral disc and can present with pain, sensory loss, muscle weakness, and functional limitations. Because the C5-T1 nerve roots provide motor and sensory innervation from the shoulder to the hand, SDH can cause not only pain but also impairments in somatosensory perception, tactile sensations, and proprioceptive awareness. Nerve root compression disrupts the integrity of sensory functions such as touch, vibration, and two-point discrimination, negatively impacting upper extremity abilities. Furthermore, pain and central sensitization processes lower the pain threshold, further limiting motor performance and activities of daily living. Therefore, the combined evaluation of somatosensory perception, pain, and functional abilities in individuals with SDH is crucial for a holistic understanding of the clinical picture.

ELIGIBILITY:
Inclusion criteria for volunteers in the study: Neck pain lasting at least 3 months, Being between the ages of 18-65 with a diagnosis of cervical disc herniation, Being able to cooperate with the applied parameters, Having good cognitive function, Being literate, Agreeing to participate in the study.

For the control group, having no complaints of neck pain and not having any neck-related diagnosis.

Exclusion criteria for volunteers in the study: Neck pain intensity during activity according to the Visual Analog Scale (VAS) below 3, Individuals who have undergone any surgery related to neck problems, Individuals who have undergone surgery related to upper extremity problems, Individuals with cervical radiculopathy, Having a systemic malignant disease anywhere in the body, Having any disease related to connective tissue or inflammatory rheumatic diseases, Having a psychiatric diagnosis and receiving treatment, Being illiterate, Not having sufficient cognitive function, Having received any neck-related physical therapy in the last 6 months for the CBA group.

Ages: 18 Years to 65 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Cervical disc herniation and healthy individuals
Sampling Method: Non-Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2025-10-24 (Actual); Primary Completion 2025-12-03 (Actual); Study Completion 2026-03-12 (Estimated)

PRIMARY OUTCOMES:
Upper extremity functionality | 24-48 hours
  Upper extremity functionality will be assessed using the Disabilities of the Arm, Shoulder, and Hand questionnaire and Purdue Pegboard Manual Dexterity Test.The total score ranges from 0 to 100, with higher scores indicating a higher level of upper extremity disability.
Pain Threshold and Tolerance Assessment | 24-48 hours
  Participants' pain threshold and tolerance to pressure are assessed using a digital algometer (JTech Medical Industries, ZEVEX Company).
Pain Assessment evaluates | 24-48 hours
  Pain Assessment evaluates the intensity of pain felt by patients in centimeters (cm) during different activities and time periods (rest, activity and night).
Somatosensory Perception Tests | 24-48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Dilan Demirtas Karaoba, Iğdır, Iğdir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No